CLINICAL TRIAL: NCT07387406
Title: A Culturally Adapted Sleep Intervention Program for Older Asian Immigrants With Limited English Proficiency
Brief Title: Sleep Learning Education and Empowerment for Older Korean Immigrants
Acronym: SLEEP-OK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Yeonsu Song, PhD, RN, FNP, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R21AG086817 (NIH); 1R21AG086817-01A1 (NIH)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Insomnia Chronic
Keywords: older Korean Americans; sleep; behavioral approach
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Intervention Program (Experimental): This is a culturally adapted sleep education program built upon key components of cognitive behavioral therapy for insomnia (CBT-I)
  Interventions: Behavioral: CBT-I based sleep intervention
- Control (Placebo Comparator): This involves with general information about sleep
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: CBT-I based sleep intervention — A multicomponent behavioral sleep program, consisting of sleep compression, stimulus control, sleep hygiene, relaxation, daily physical activity, and light exposure
  Arms: Sleep Intervention Program
Behavioral: Sleep Education — This group will receive information about sleep and aging, but without specific or individualized recommendations
  Arms: Control

SUMMARY:
Poor sleep is common among Asian Americans. Untreated sleep problems increase the risk of chronic diseases, cognitive decline, and mortality. Cognitive behavioral therapy for insomnia (CBTI) is considered the first-line treatment for chronic sleep problems and has demonstrated significant improvement in sleep health among older adults. However, existing CBTI is built upon Western culture, making it challenging to apply for Asian immigrants who maintain close ties to their native cultures that shape and influence their sleep habits. Addressing the lack of availability of a culturally adapted sleep intervention program is the first step to filling the gap in sleep health disparity among Asian immigrants.

This study aims to pilot test the feasibility and the preliminary efficacy of a culturally adapted sleep intervention program among older Korean immigrants with poor sleep, one of the fastest-growing immigrant groups in the United States with limited access to mainstream sleep therapies.

DETAILED DESCRIPTION:
Poor sleep is common among Asian Americans. Untreated sleep problems increase the risk of chronic diseases, cognitive decline, and mortality. Addressing the lack of availability of a culturally adapted sleep intervention program is the first step to filling the gap in sleep health disparity among Asian immigrants. This study aims to evaluate its feasibility and preliminary efficacy of a culturally adapted sleep education program ("SLEEP-OK") in a pilot randomized clinical trial. Study participant (N=32) will be randomized to either our culturally adapted, manual-based sleep intervention group (n=16) or the information-only control group (n=16) at our community partner serving older Korean immigrants. The study will evaluate the feasibility of the intervention and the preliminary effects of the intervention on sleep health outcomes among Korean immigrants at baseline and post-intervention (i.e., immediately after the last session of the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Korean immigrants (i.e., being a resident of the United States with a birthplace in Korea)
* Able to speak, read, and write in Korean
* Aged at least 60 years
* Have a score of at least 15 on a Korean version of the Insomnia Severity Index
* Able to ambulate with or without an assistive device
* Have a score of at least 23 on a Korean version of the Montreal Cognitive Assessment (MoCA)
* Score less than 5 on STOP-BANG (or proceed with an additional testing [Watch Peripheral Arterial Tonometry (WatchPAT) and the Epworth Sleepiness Scale if score is equal to or greater than 5 on STOP-BANG)

Exclusion Criteria:

* Those who are bedbound
* Those who do not meet the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for insomnia disorder
* Those who have an untreated apnea-hypopnea index (AHI) at least 15 (moderate obstructive sleep apnea) and Epworth Sleepiness Scale (ESS) at least 11 (indicating mild sleepiness) OR AHI is equal to or greater than 30 (irrespective of ESS)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Objective Sleep Efficiency | Immediately after the last session of the intervention
  Nighttime sleep efficiency (i.e., mean percent of time in bed spent asleep at nighttime) will be calculated from 7 consecutive days and nights of wrist actigraphy (Scores range from 0 to 100%, with higher values indicating better objective sleep quality)
Subjective Sleep Quality | Immediately after the last session of the intervention
  Total score on the Korean version of the Insomnia Severity Index (ISI) will be used as a measure of subjective sleep (Scores range from o to 18, with lower values indicating better subjective sleep quality)

SECONDARY OUTCOMES:
Acceptability of the Intervention | Immediately after the last session of the intervention
  Focus group interviews will be conducted to collect the benefits and challenges of following the sleep intervention program

OTHER OUTCOMES:
Feasibility of Recruitment | Immediately after enrolled
  The number of participants approached who agreed to participate will be measured
Feasibility of Randomization and Retention | Immediately after enrolled
  The number of participants lost at a post-treatment assessment will be measured
Adherence to the Intervention | Immediately after the last session of the intervention
  The total number of sessions and the percentage of days that participants met goals for recommendations throughout the intervention program will be measured
Interventionist Adherence | Immediately after the last session of the intervention
  The percentage of completion of delivery of each component in sessions throughout the intervention program will be measured

IPD SHARING:
Plan to Share IPD: Yes
IPD difficulty masking the identity of participants will not be shared publicly. However, all de-identified data and metadata will be made available through National Sleep Research Resource (NSRR), an NHLBI-funded resource at the time of the associated publication or the end of this project year, whichever comes first. Final research data and metadata will be shared by the end of the project period or at the time of publication, whichever is sooner, and will remain accessible indefinitely.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: by the end of the project period or at the time of publication, whichever is sooner,